CLINICAL TRIAL: NCT01084681
Title: Multicenter Randomized Trial on Selective Endovascular Aneurysm Occlusion With Coils Versus Parent Vessel Reconstruction Using the SILK Flow Diverter (MARCO POLO Post-Market Clinical Investigation)
Brief Title: Efficacy Trial of Intracranial Aneurysm Treatment Using Two Different Endovascular Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Balt International (Industry)
Responsible Party: Linda Nicolini / Director of Market Development, Balt International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Balt 2010-01
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Intracranial Aneurysms
Keywords: SILK flow diverter, intracranial stents, intracranial aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILK Artery Reconstruction Device (Active Comparator): One arm will receive only the commercially available SILK Artery Reconstruction Device [flow diverter] (no intracranial coils are to be used in association with the SILK device).
  Interventions: Device: Endovascular treatment of intracranial aneurysms
- Coils (Active Comparator): The other arm will be treated with commercially available intracranial coils: the coils can be used with eventual balloon remodeling and/or stents when necessary.
  Interventions: Device: Endovascular treatment of intracranial aneurysm with coils

INTERVENTIONS:
Device: Endovascular treatment of intracranial aneurysms — Endovascular treatment with the SILK Artery Reconstruction Device for occluding intracranial aneurysms.
  Arms: SILK Artery Reconstruction Device
Device: Endovascular treatment of intracranial aneurysm with coils — Endovascular treatment with commercially available intracranial coils for occluding intracranial aneurysms.
  Other Names: Endovascular treatment of intracranial aneurysms
  Arms: Coils

SUMMARY:
To date the standard non-surgical treatment strategy for treating un-ruptured intracranial aneurysms is the use of either coils or self-expandable stents. This post-market clinical investigation compares the efficacy of using the CE-marked, commercially available SILK Artery Reconstruction Device against commercially available intracranial coils in the endovascular treatment (occlusion) of intracranial aneurysms.

DETAILED DESCRIPTION:
To date the standard non-surgical treatment strategy for treating un-ruptured intracranial aneurysms is the use of either coils or self-expandable stents. The flow diverter stent concept is based upon the hemodynamic exclusion of the aneurysm sac, without coils being eventually placed within the sac. The primary objective of this post-market clinical investigation is to demonstrate that when using the CE-marked, commercially available SILK Artery Reconstruction Device in the indication for which it is approved, notably for the treatment (occlusion) of intracranial aneurysms, the anatomical results are superior compared to standard treatment with commercially available intracranial coils (used with eventual balloon remodeling and/or stents when necessary). It is a prospective, randomized, unblinded, multi-center post-market clinical investigation. The patient population comprises a maximum of 160 subjects with at least one documented untreated, unruptured intracranial aneurysm suitable for occlusion with an intracranial device. Subject enrollment will require a maximum of 18 months. Enrolled subjects will be followed for 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least one documented untreated, unruptured intracranial aneurysm
* The intracranial aneurysm is non-thrombosed and non-hemorrhagic
* Saccular Carotid Siphon: with a sac diameter of ≥7mm to ≤15mm
* Lateral vertebral aneurysms of V4, and side-wall basilar trunk aneurysms
* Target aneurysm morphology permits the use of intracranial devices, as determined by the treating physician
* Subject greater than or equal to 18 years old
* Life expectancy greater than or equal to 12 months
* Subject (or subject's legally authorized representative) has provided written informed consent
* Subject is willing and able to comply with protocol follow-up requirements

Exclusion Criteria:

* Subject is under guardianship
* Significant atherosclerotic disease, stenosis, tortuosity or other condition preventing microcatheter access to the target aneurysm(s)
* Vessel branch arising from the aneurysm sac
* Fusiform aneurysm
* Ruptured aneurysm
* Bifurcation aneurysms (MCA, ACoA)
* Recurrent aneurysm
* Presence of an intracranial stent on the side that is to be treated
* High risk surgical subjects with significant pre-existing co-morbid condition(s), not treated or well controlled with standard therapy
* Bleeding disorder which would preclude percutaneous intervention and/or anti-thrombotic therapy; resistance to anti-platelet treatment
* Intracranial intervention performed within 30 days prior to the procedure or elective intracranial intervention planned within 12 months following the procedure
* Major surgical procedure (e.g., coronary artery bypass graft, valve replacement, abdominal aortic aneurysm repair, bowel resection) performed within 30 days preceding or planned within 12 months following the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 12 months
  The primary objective is to demonstrate that when using the SILK Artery Reconstruction Device in the indication for which it is approved, notably for the treatment (occlusion) of intracranial aneurysms, the anatomical results are superior compared to standard treatment with commercially available intracranial coils. Therefore, angiographic assessment will measure efficacy by determining the percentage of subjects in each of the two arms experiencing complete occlusion of the aneurysm at 12 months post-procedure.

SECONDARY OUTCOMES:
Safety | 12 months
  Safety will be evaluated as follows:
  1. Peri-procedural ischemic and hemorrhagic adverse events
  2. Peri-procedural technical complications
  3. Death from any cause
  4. Neurological deterioration
  5. Cranial nerve deficit
  6. General adverse events
  In addition, Subject Quality of Life (QOL) will be measured at baseline and at 12 months post-procedure using the EuroQol questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Moret, MD, Study Chair — Beaujon Hospital - Paris Diderot University (Paris, France)
Locations (1):
- Universitätsklinikum Würzburg; Abteilung für Neuroradiologie, Würzburg, Germany